NCT01996605

Official Title: Efficacy of Intrathecal Oxytocin in Human Volunteers

IRB-Approved Date: 1/25/22



Department/Section of Anesthesiology

## EFFICACY OF SPINAL OXYTOCIN IN HUMAN SUBJECTS

Informed Consent Form to Participate in Research James C. Eisenach, M.D., Principal Investigator

#### Introduction

You are invited to be in a research study. Research studies are designed to gain scientific knowledge that may help other people in the future. You are being asked to take part in this study because you are a healthy subject. Your participation is voluntary. Please take your time in making your decision as to whether or not you wish to participate. Ask your study doctor or the study staff to explain any words or information contained in this informed consent document that you do not understand. You may also discuss the study with your friends and family.

# WHY IS THIS STUDY BEING DONE?

This research study is being done because pain is a significant problem for patients with a variety of medical problems and following surgery or traumatic injury. Currently available pain medications may not treat all types of pain or may treat pain only at doses that produce side effects and complications. The medication in this study may have a role in better treatment of pain. Oxytocin is commonly given by IV (into a vein) to treat certain types of pain. This is the second study in the United States to examine the effects of oxytocin given into the spinal fluid in the back. We believe that spinal oxytocin may prove to be an excellent pain killer for certain types of pain which sometimes occur with cancer or follow nerve injury after accidents or surgery. At present, there are not good treatments for this type of pain and your participation in this study may help researchers better understand this type of pain and perhaps develop new ways of treating this pain.

The goals of this study are to see if a dose of oxytocin, given into the fluid in your back near the spine has any effect on pain or discomfort in the skin sensation that will take place after applying capsaicin (chili pepper) cream. The sunburn-like sensation that people experience after having capsaicin cream applied is similar to, but much milder than, the pain that some people have after surgery and after certain types of nerve injuries.

Oxytocin has been approved by the US Food and Drug Administration (FDA), but the preparation and route of administration being used in this study has not been approved. However, the study is being conducted under the review of the FDA. At this time, there is not a form of Oxytocin that is available on the open market for spinal administration.

 Adult Consent Form

Version: 1/25/2022

In this study oxytocin will be compared to placebo. A placebo is a substance, like a sugar pill, that is not thought to have any effect on diseases or medical conditions. In this study you will either receive the active study medication, oxytocin or placebo which is not active. Placebos are used in research studies to see if the drug being studied really does have an effect

# HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

We will study 36 people at people at this research site. In order to identify the 36 subjects needed, we may need to screen as many as 40 people because some people will not qualify to be included in the study.

# WHAT IS INVOLVED IN THE STUDY?

You will have three visits (detailed below) to the Clinical Research Unit (CRU). If you take part in this study, all of the test and procedures performed will be solely for research purposes.

You will be randomized into one of the study groups described below. Randomization means that you are put into a group by chance. It is like flipping a coin. You will have a one in three chance of being placed in any group.

Group 1- will receive 15 micrograms of spinal oxytocin

Group 2- will receive 150 micrograms of spinal oxytocin

Group 3- will receive saline (placebo) in the spinal injection

Neither you nor the investigator will know which group you are in. This is done so that a fair evaluation of results can be made. This information is available to the researchers if needed in an emergency.

If you take part in this study, you will have the following tests and procedures:

## **PROCEDURES**

<u>Vital Signs</u>: we will monitor your blood pressure, heart rate and oxygen saturation (amount of oxygen in your blood).

**Electrocardiogram (EKG):** tracing of the rhythm of your heart.

<u>Laboratory Testing</u>: female participants of child-bearing potential will have blood drawn to determine that they are not pregnant.

Thermal Heat Testing: we will train you to accurately describe pain from a small heat probe (1.5 inches). The tip of the heat probe that will be applied to you're the skin on your forearm is about the size of a penny. The thermal heat probe will be controlled by a computer that is programmed to deliver temperatures that range from skin temperature up to a temperature that is hot (124 °F) and uncomfortable, but does not burn your skin. We will ask you to rate the pain by using a sliding scale. Most volunteers find that they can learn to tell very small

 Adult Consent Form

differences in the temperature probe accurately.

**Light Touch Testing:** a von Frey filament (a plastic thread like a paint brush bristle) and a cotton wisp (Q-tip) will be lightly applied to your skin. We will ask you to tell us when you feel a difference in the sensitivity on your skin. We will use a washable marker to "mark" the areas that you tell us are more sensitive.

<u>Capsaicin Testing</u>: we will place the thermal heat probe on your calf and warm the area to a temperature of 113°F for 5 minutes. During this five minute warming period we will ask you to give a pain rating each minute for any pain you are experiencing. We will then test your skin sensations with the filament and cotton wisp, after which *capsaicin cream (an over-the-counter pain relief cream)* will be put on your skin in the same spot as the heat probe. The cream will be on your skin for 30 minutes. During this time we will ask you to rate any pain you feel every 5 minutes. We will remove the capsaicin cream from your skin with a soft cloth. After removing the cream, we will then test your skin sensations with the filament and Q-tip as described in the Light Tough Testing.

**'Rekindling' of the Capsaicin Testing Area**: 40 minutes after removing the capsaicin cream, we will apply thermal heat at a temperature of 104°F to the same area where the capsaicin cream was applied to. We will leave the heat on your skin for five minutes. At the end of the five minutes we will ask you to rate any pain you are experiencing. This procedure is known as "rekindling". We will test your skin sensations with the filament and cotton wisp (Light Touch Testing) before and after this second heating.

**Blood Draw:** we will draw 3 blood samples from the IV that we have placed in your arm; the total amount for each sample will be 1 teaspoon. We will draw a total of 3 teaspoons. If we cannot draw the blood from your IV we will perform an additional venipuncture.

#### **Study Visit 1:**

During the first study visit we will record your we will measure your blood pressure, heart rate, and we will place a clip on your finger which will measure the oxygen in your blood. We will perform an electrocardiogram (EKG), to obtain a baseline tracing of your heart and female participants of child-bearing potential will have approximately 1 teaspoon of blood drawn for a pregnancy test. We will also train you to rate pain in response to heat applied to your forearm and the outside of your lower leg (Thermal heat testing and Capsaicin testing). We will then perform one cycle of the capsaicin testing, providing you the opportunity to experience the testing and to be trained in evaluating the area of sensitivity. This visit will last approximately 2 hours

#### **Study Visit 2:**

On the morning of the second session you will come to the Clinical Research Center (CRU) having had nothing to eat or drink after midnight. We will record your blood pressure, heart rate, the amount of oxygen in your blood, and we will connect you to a heart monitor. We will again perform a short training session with the heat probe. Then we will insert an intravenous catheter into a vein in your arm and you will get IV fluid through this catheter.

Page **3** of **12** Adult Consent Form

We will then ask you to curl up into a ball on your side on a bed and put a spinal needle into the spinal space in the lowest part of your back after numbing the skin with lidocaine. After successfully placing the spinal needle, we will take a sample approximately one-half of a teaspoon of your spinal fluid and then we will then inject the oxytocin or placebo according to the randomization that has been selected for you. The spinal needle will then be withdrawn and you will be asked to lie on your back with the head of the bed elevated slightly.

Thirty minutes after the spinal injection we will perform the testing with the capsaicin cream. We will perform 3 cycles of testing on the area where the capsaicin was applied at 40 minute intervals.

Multiple times during this day (from just before the spinal until 3.5 hours after the spinal injection) we will measure your blood pressure, measure the oxygen in your bloodstream with the finger-clip, examine you to test your arm and leg strength, and sensations, (to test for any changes in the strength or sensation you have in your arms and legs) and ask you to about any other sensations you may be experiencing. We will also monitor your electrocardiogram throughout the study period.

About 3.5 hours after the spinal injection we will stop gathering information for the study. To go home, you must not have any side effects that would prevent you from walking (like dizziness, unsteadiness). You must have someone drive you home and you must be available for us to call you at home. We will call you 6 hours after the spinal drug injection and 12 hours after the spinal drug injection. You must call us if you have any questions or concerns during this period. There is a remote chance that should you experience side effects which are concerning, we will keep you in the hospital overnight.

#### **Study Visit 3:**

Version: 1/25/2022

You must return to the CRU approximately 24 hours after the spinal drug injection. You will have approximately 1 teaspoon of blood withdrawn from a vein during the 24 hour follow up visit to have your electrolytes evaluated. After all of the measurements are finished, the study will be complete. We will call you daily for 5 days, then weekly for 1 month, then approximately 6 months after the study and ask you about any symptoms that you believe you might have experienced. If at any time you have a question or a concern, please call us.

# Storage of Biological Tissue

If you agree to participate in this study, we will draw one-half of a teaspoon (2 milliliters) of cerebrospinal fluid (CSF) prior to injection of the study medication to use for future research. This sample will be kept and may be used in future research to learn more about other diseases. Your sample will be obtained in the Clinical Research Unit by the Anesthesiology Department at Wake Forest University Baptist Medical Center. The sample will be stored in the Pain Mechanisms Laboratory and it will be given only to researchers approved by Dr. James Eisenach. An Institutional Review Board (IRB) must also approve any future research study using your tissue sample. In order to participate in this study, you must be willing to provide this sample for future research.

Your CSF sample will be stored with a unique identifier and will not include any identifiable

 Adult Consent Form

information about you such as your name, address, telephone number, social security number, medical record number or any of the identifiers outlined in the HIPAA Privacy Rule. The unique identifier will be a randomly assigned number and only the principal investigator will have access to the code that links the unique identifier to you. Your name, address, social security number, etc., will never be disclosed to future researchers and neither will the code that links your identifiers to the sample.

The research that may be performed with your CSF sample is not designed to help you specifically. There is no personal benefit to you from taking part in this aspect of the research study. It might help people who have diseases at some point in the future, but it is not known if this will happen. The results of the research performed with your CSF will not be given to you or your doctor. The results will not be put in your medical record. The research using your CSF sample will not affect your care.

Your CSF sample will be used only for research and will not be sold. The findings from this research may result in the future development of products that are of commercial value. There are no plans to share any of the profits with you which may occur as a result of the research.

# HOW LONG WILL I BE IN THE STUDY?

You will attend 3 study visits. Following visit 2, we will contact you by telephone 6 and 12 hours following the spinal drug injection. Following visit 3, we will contact you by telephone daily for 5 days, then weekly for 1 month, then approximately 6 months later. Total study duration is approximately 6 months.

You can stop participating at any time.

# WHAT ARE THE RISKS OF THE STUDY?

Being in this study involves some risk to you. The risks are given below. You should discuss the risk of being in this study with the study staff.

#### **Heat Probe**

You may experience brief pain during the thermal heat testing.

#### Capsaicin

Risks of the capsaicin include: pain and allergic reaction.

# Oxytocin

The safety of spinal oxytocin has been extensively examined in animals, with no evidence of any nerve damage or other lasting effects, the FDA has approved this investigational study for humans, and nearly 1000 humans have received spinal oxytocin in China without reported problems. Although this all suggests that it is safe to administer oxytocin, the exact risks are unknown. We will monitor you for many theoretical problems such as your level of sleepiness, changes in your blood pressure, how fast your heart is beating, and your urge to breathe. We will treat any side effects that you may experience if the changes are enough to concern us.

Page **5** of **12** Adult Consent Form

#### **Spinal Procedures**

Risks associated with the spinal procedures are mild bruising and soreness in the area. There is a risk (less than 1%) of developing a headache from the spinal needles. If you develop a headache that does not go away and is bothersome, we will talk to you about an epidural blood patch. This is a simple procedure, which would involve putting a needle in the epidural space in your back and injecting some blood taken from your arm. This procedure is 95% (95 times out of 100) effective in treating the headache. However you would have a 1 in 3 chance of having a backache for a few days. Rarely (5 out of 100 times) is a 2nd blood patch needed. Other risks of the epidural blood patch are the same as the spinal. You will not be charged if you need an epidural blood patch to treat a headache. The risk of paralysis, infection or nerve damage from a spinal procedure is extremely rare, less than one chance in 20,000. The numbing medicine that we put under your skin right before the spinal needle is inserted may cause you to have a brief period (about 5 seconds) of mild discomfort.

We may be unable to place the spinal needles due to the shape of your back. If we cannot place the spinal needles, you would no longer be able to continue participating in the study. You will be paid as detailed below.

#### **Risks from Needle Insertions**

You may experience discomfort, bruising and/or bleeding where the needle is inserted. Occasionally some people become dizzy lightheaded or feel faint. Infection may occur on rare occasions.

## For Electrocardiogram (ECG):

The electrode pads used during the ECG may cause minor skin redness or irritation.

You can call the study staff at any time if you think you might be having any of the side effects discussed above. Also, the study staff will be telephoning you each day for 5 days after the study, then weekly for 1 month, then approximately 6 months after the study and ask you about any symptoms that you believe you might have experienced. If at any time you have a question or a concern, please call us.

In addition, there is a slight risk of a breach of confidentiality. We will do our best to protect your confidential information. There also may be other side effects that we cannot predict. You should tell the research staff about all the medications, vitamins and supplements you take and any medical conditions you have. This may help avoid side effects, interactions and other risks.

Taking part in this research study may involve providing information that you consider confidential or private. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe.

A Data Safety and Monitoring Committee, an independent group of experts, will be reviewing the data from this research throughout the study.

 Adult Consent Form

# Reproductive Risks and other Issues to Participating in Research

Pregnant women are excluded from participation in this study. Because some methods of birth control are not 100% reliable, a pregnancy test is required at least 10 days from your last normal menstrual period, if you are a sexually active woman of childbearing potential.

# ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

You are not expected to receive any direct benefit from taking part in this research study. We hope the information learned from this study will benefit other people in the future.

# WHAT OTHER CHOICES ARE THERE?

This is not a treatment study. Your alternative is to not participate in this study.

# WHAT ABOUT MY HEALTH INFORMATION?

Your personal health information and information that identifies you ("your health information") may be given to others during and after the study. This is for reasons such as to carry out the study, to determine the results of the study, to make sure the study is being done correctly, to provide required reports and to get approval for new products.

Some of the people, agencies and businesses that may receive and use your health information are the research sponsor; representatives of the sponsor assisting with the research; investigators at other sites who are assisting with the research; central laboratories, reading centers or analysis centers; the Institutional Review Board; representatives of Wake Forest University Health Sciences and North Carolina Baptist Hospital; representatives from government agencies such as the Food and Drug Administration (FDA), the Department of Health and Human Services (DHHS) and similar agencies in other countries.

Some of these people, agencies and businesses may further disclose your health information. If disclosed by them, your health information may no longer be covered by federal or state privacy regulations. Your health information may be disclosed if required by law. Your health information may be used to create information that does not directly identify you. This information may be used by other researchers. You will not be directly identified in any publication or presentation that may result from this study unless there are photographs or recorded media which are identifiable.

- Monitors, auditors, IRB or other regulatory agencies will be granted direct access to the
  participant's original medical record for verification of clinical trial procedures or data,
  without violating confidentiality of the participant and to the extent permitted by other
  applicable laws.
- 2) Representatives from government agencies such as the US Food and Drug Administration (FDA), the Department of Health and Human Services (DHHS).
- 3) Representatives from government agencies such as the Office for Human Research Protections and other similar agencies.

 Adult Consent Form

Version: 1/25/2022

If required by law or court order, we might also have to share your Protected Health Information with a judge, law enforcement officer, government agencies, or others. If your Protected Health Information is shared with any of these groups it may no longer be protected by federal or state privacy rules.

Any Protected Health Information collected from you in this study that is maintained in the research records will be kept for an indeterminate period of time. This authorization does not expire and any research information entered into your medical record will be kept for as long as your medical record is kept by the Medical Center. You will not be able to obtain a copy of your Protected Health Information in the research records until all activities in the study are completely finished

You can tell Dr. James C. Eisenach that you want to take away your permission to use and share your Protected Health Information at any time by sending a letter to this address:



Version: 1/25/2022

However, if you take away permission to use your Protected Health Information you will not be able to be in the study any longer. We will stop collecting any more information about you, but any information we have already collected can still be used for the purposes of the research study.

By signing this form you give us permission to use your Protected Health Information for this study.

If you choose to participate in this study, your medical record at Wake Forest University Baptist Medical Center will indicate that you are enrolled in a clinical trial. Information about the research and any medications or devices you are being given as a participant may also be included in your medical record. This part of the medical record will only be available to people who have authorized access to your medical record. If you are not a patient at this Medical Center, a medical record will be created for you anyway to ensure that this important information is available to doctors in case of an emergency.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this Web site at any time.

Laboratory test results and other medical reports created as a result of your participation in the research study may be entered into the computer systems of Wake Forest University Health Sciences and North Carolina Baptist Hospital. These will be kept secure, with access to this information limited to individuals with proper authority, but who may not be directly involved

 Adult Consent Form with this research study.

A North Carolina Baptist Hospital (NCBH) medical record will be created for all study participants. Information about your participation in the study will be placed in the NCBH medical record, along with any routine medical test results that were obtained at NCBH as part of this study.

# WHAT ARE THE COSTS?

There are no costs to you for taking part in this study. All study costs, including any study medications and procedures related directly to the study, will be paid for by the study. Costs for your regular medical care, which are not related to this study, will be your own responsibility.

# WILL YOU BE PAID FOR PARTICIPATING?

You will be paid \$500(outlined below) if you complete all the scheduled study visits. If you withdraw for any reason from the study before completion you will be paid for the portion of the study that you completed.

- Placement of IV: \$25
- Placement of Spinal: \$125 and study drug administration (if spinal placement is unsuccessful, the study will be abandoned and the subject paid for the portion completed)
- Application of capsaicin cream: \$25 for each application (total \$50)
- Completion of entire study (completing 3 study visits with all data collection): \$300

To receive payment, you must provide your social security number, name and address so that we can comply with IRS (Internal Revenue Service) reporting requirements. When payments are reported to the IRS we do not let them know what the payment is for, only that you have been paid. If you do not wish to provide this information you can still take part in this study but you will not be paid.

The findings from this research may result in the future development of products that are of commercial value. There are no plans to provide you with financial compensation or for you to share in any profits if this should occur.

#### WHO IS SPONSORING THIS STUDY?

This study is being sponsored by the National Institutes of Health. The sponsor is providing money or other support to Wake Forest University Health Sciences to help conduct this study. The researchers do not, however, hold a direct financial interest in the sponsor or the product being studied.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires

 Adult Consent Form

disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects. The Certificate cannot be used to refuse a request for information from personnel of the United States federal or state government agency sponsoring the project that is needed for auditing or program evaluation by The National Institute of Health which is funding this project or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). You should understand that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it

# WHAT HAPPENS IF YOU EXPERIENCE AN INJURY OR ILLNESS AS A RESULT OF PARTICIPATING IN THIS STUDY?

Should you experience a physical injury or illness as a direct result of your participation in this study, Wake Forest University School of Medicine maintains limited research insurance coverage for the usual and customary medical fees for reasonable and necessary treatment of such injuries or illnesses. To the extent research insurance coverage is available under this policy the reasonable costs of these necessary medical services will be paid, up to a maximum of \$25,000. Wake Forest University Baptist Medical Center holds the insurance policy for this coverage. It provides a maximum of \$25,000 coverage for each claim and is limited to a total of \$250,000 for all claims in any one year. The Wake Forest University School of Medicine, and the North Carolina Baptist Hospitals, Incorporated do not assume responsibility to pay for these medical services or to provide any other compensation for such injury or illness. Additional information may be obtained from the Medical Center's Director of Risk and Insurance Management, at

If you are injured, the insurer may require information such as your name, social security number, and date of birth in order to pay for your care. This is because the insurer is required by law to report any payments made to cover the care of any persons who are members of a government insurance plan to the Department of Health and Human Services.

You do not give up any legal rights as a research participant by signing this consent form. For more information on medical treatment for research related injuries or to report a study related illness, adverse event, or injury you should call Dr. James Eisenach at hours you should call the study coordinator by calling

# WHAT ARE MY RIGHTS AS A RESEARCH STUDY PARTICIPANT?

Taking part in this study is voluntary. You may choose not to take part or you may leave the study at any time. Refusing to participate or leaving the study will not result in any penalty or loss of benefits to which you are entitled. If you decide to stop participating in the study we encourage you to talk to the investigators or study staff first to learn about any potential health or safety consequences. The investigators also have the right to stop your participation in the study

 Adult Consent Form

at any time. This could be because you failed to follow instructions or because the entire study has been stopped.

You will be given any new information we become aware of that would affect your willingness to continue to participate in the study.

This study will be enrolling students from the Wake Forest University and Wake Forest University Medical Center campus. In addition to your rights as a research participant noted in the previous section, as a student, you are under no obligation to participate in this study. You may refuse to participate or withdraw from the study at any time and for any reason without affecting your grades, performance evaluations, or assignments. You will not be pressured into participating in this research study by any statements or implied statements that your grades, performance evaluations or assignments will be affected by your willingness to enroll in the study. Your medical records/information will not be used by the faculty, administration or study staff to make decisions regarding the status of your medical benefits. If you have questions regarding your enrollment in the study and your status as a medical student, please contact the Office of Student Services for additional information.

# WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

| For questions about the study or in the | event of a research-related injury, contact the study |
|---|---|
| investigator, Dr. James Eisenach at | or after hours you should page the study |
| coordinator by calling | |

The Institutional Review Board (IRB) is a group of people who review the research to protect your rights. If you have a question about your rights as a research participant, or you would like to discuss problems or concerns, have questions or want to offer input, or you want to obtain additional information, you should contact the Chairman of the IRB at

You will be given a copy of this signed consent form.

#### SIGNATURES

Version: 1/25/2022

I agree to take part in this study. I authorize the use and disclosure of my health information as described in this consent and authorization form. If I have not already received a copy of the Privacy Notice, I may request one or one will be made available to me. I have had a chance to ask questions about being in this study and have those questions answered. By signing this consent and authorization form, I am not releasing or agreeing to release the investigator, the sponsor, the institution or its agents from liability for negligence.

| Subject Name (Printed): | | | |
|-------------------------|-------|--------|-------|
| Subject Signature: | Date: | Time: | am pn |
| Subject Signature: | Date: | i ime: | am |

 Adult Consent Form

| Person Obtaining Consent: | Date: | Time: | am pm |
|---------------------------|-------|-------|-------|

Version: 1/25/2022